CLINICAL TRIAL: NCT03617471
Title: Pharmacokinetic Study of Paracetamol in Patients Over 80 Years Hospitalized to an Acute Geriatric Ward
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Principal Investigator, Isabelle Spriet, PharmD, PhD, Universitaire Ziekenhuizen KU Leuven
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: S58396 - mp05485
Record Dates: First submitted 2016-11-29; First posted 2018-08-06 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paracetamol oral tablets 1g tid (Experimental): Patients received paracetamol one gram three times daily. Venopuncture for PK profiling
  Interventions: Procedure: Venopuncture for PK profiling
- Paracetamol oral granules 1g tid (Experimental): Patients received paracetamol one gram three times daily. Venopuncture for PK profiling
  Interventions: Procedure: Venopuncture for PK profiling

INTERVENTIONS:
Procedure: Venopuncture for PK profiling — Blood samples at T0, T0.5, T1, T2, T4, T6
  Other Names: Blood sampling for paracetamol dosage

SUMMARY:
The goal of this exploratory study is the characterization of the pharmacokinetic (PK) profile of paracetamol in older patients and the specific PK (pharmacokinetic) variables associated with plasma exposure in this population.

DETAILED DESCRIPTION:
The goal of this exploratory study is the characterization of the pharmacokinetic profile of paracetamol in older patients and the specific PK variables associated with plasma exposure in this population. The primary endpoint is the identification of the pharmacokinetic parameters: area under the curve (AUC), peak plasma concentration after administration of paracetamol (Cmax) and the time at which the Cmax is observed (Tmax) of paracetamol. The secondary endpoint consists of 3 sub-endpoints:

1. The variability in plasma exposure: volume of distribution (Vd), clearance (Cl) and elimination half-life (t1/2)
2. The association between the PK parameters and pathophysiological factors
3. The correlation between PK parameters and clinical parameters.

ELIGIBILITY:
Inclusion Criteria:

* a minimum age of 80 years
* admission to the acute geriatrics ward
* oral intake of paracetamol 1000 milligram (mg) in tablet form tid
* a steady state situation (defined as at least 4 consecutive intakes of paracetamol before sampling)

Exclusion Criteria:

* palliative care setting with downgrading of care

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-11; Primary Completion 2016-01 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Identification of the pharmacokinetic parameters: AUC | 8 hours (= during 1 dosing interval at steady state)
  Area under the curve (AUC)
Identification of the pharmacokinetic parameters: Cmax | 8 hours (= during 1 dosing interval at steady state)
  Peak plasma concentration after administration of paracetamol (Cmax)
Identification of the pharmacokinetic parameters: Tmax | 8 hours (= during 1 dosing interval at steady state)
  The time at which the Cmax is observed (Tmax) of paracetamol

SECONDARY OUTCOMES:
Variability in plasma exposure: Vd | 8 hours (= during 1 dosing interval at steady state)
  Volume of distribution (Vd)
Variability in plasma exposure: t1/2 | 8 hours (= during 1 dosing interval at steady state)
  Elimination half-life (t1/2)
Variability in plasma exposure: Cl | 8 hours (= during 1 dosing interval at steady state)
  Clearance (Cl)
The association between the AUC (area under the curve) of paracetamol and patient related factors. | 8 hours (= during 1 dosing interval at steady state)
  Multivariate analysis will be performed with AUC (area under the curve) as outcome. This will allow to identify variables influencing AUC of paracetamol. Patient related factors include amongst others age, weight, albumin, bilirubin, serum creatinin and co medication.
The association between the AUC (area under the curve) of paracetamol and pain scores. | 8 hours (= during 1 dosing interval at steady state)
  Pain scores will be based on the Numeric Rating Scale with a score of 0 indicating no pain and a score of 10 indicating worst imaginable pain.
Correlation between immuno assay method and the Liquid chromatography-tandem mass spectrometry (LC-MS/MS) method to determine paracetamol concentrations in serum | 8 hours (= during 1 dosing interval at steady state)
  Correlation between two different assays will be determined through Bland Altman statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Spriet, PharmD PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Universitaire Ziekenhuizen Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No